CLINICAL TRIAL: NCT06733168
Title: The Impact of PEEP-guided Electrical Impedance Tomography on Oxygenation and Pulmonary Mechanics in Moderate-to-severe ARDS
Acronym: PEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam Military Medical University (Other)
Collaborators: Hanoi Medical University (Other); Bach Mai Hospital (Other)
Responsible Party: Principal Investigator, Nguyen Dang Thu, PhD, MD, Vietnam Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TrungHSTC 5532/BM-HDDD
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Syndrome Distress; Positive End-Expiratory Pressure; Mechanical Ventilation; Electrical Impedance Tomography (EIT)
Keywords: Acute respiratory syndrome distress; Mechanical Ventilation; Positive End-Expiratory Pressure; electrical impedance tomography; blood oxygenation; pulmonary mechanics
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, single center, ramdomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT-PEEP setting (Active Comparator): Patients will have PEEP settings determined by EIT guidance following a stepwise decremental PEEP trial
  Interventions: Device: electrical impedance tomography
- ARDSNet-PEEP setting (Placebo Comparator): PEEP will be adjusted using the low FiO2-PEEP table to achieve oxygenation targets: SpO2 between 88% and 95% and PaO2 between 55 mmHg and 80 mmHg
  Interventions: Other: Non-EIT

INTERVENTIONS:
Device: electrical impedance tomography — Before initiating recruitment maneuver, all patients were placed on mechanical ventilation set according to the ARDSnetwork strategy for 10 minutes, ensuring SpO2 of 88-95%, PaO2 of 55-80 mmHg, and a mean arterial pressure (MAP) ≥ 65 mmHg.
  * PEEP was incrementally increased by 5 cmH2O every minute: from 10 to 15, to 20, and finally to 25 cmH2O, with a maximum pressure limit of 40 cmH2O.
  * Following recruitment maneuver at the final PEEP level, the process of identifying the optimal PEEP was initiated.
  * Then, PEEP will be set to 20 cmH2O and was gradually decreased by 2 cmH2O every 30 seconds until it reached 6 cmH2O or SpO2 dropped to ≤ 80%.
  * Selection of optimal PEEP: The optimal PEEP was defined as the intersection point between the alveolar overdistension and collapse curves as measured by the EIT system.
  Arms: EIT-PEEP setting
Other: Non-EIT — Patients will have PEEP set using the low FiO2-PEEP table, based on the ARDSnet protocol
  Arms: ARDSNet-PEEP setting

SUMMARY:
Acute respiratory distress syndrome (ARDS) in its moderate to severe forms is associated with high mortality. Mechanical ventilation (MV) remains the cornerstone of ARDS management but carries a significant risk of ventilator-induced lung injury (VILI). Positive end-expiratory pressure (PEEP), a fundamental component of MV, is widely utilized in clinical practice; however, optimal PEEP selection for patients with moderate to severe ARDS remains a complex and unresolved challenge. Electrical impedance tomography (EIT), a bedside imaging modality that evaluates regional ventilation distribution, offers a means of individualizing PEEP settings in mechanically ventilated patients. By balancing the competing risks of alveolar overdistension and collapse, EIT facilitates precision in PEEP titration. This study compares the impact of EIT-guided PEEP selection versus the conventional low FiO2-PEEP table on blood oxygenation and pulmonary mechanics.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled trial designed to evaluate the effects of PEEP settings guided by electrical impedance tomography (EIT) on clinical outcomes in patients with moderate to severe ARDS undergoing lung-protective ventilation. Adult intubated patients with moderate to severe ARDS will be enrolled in the study.

Patients in the intervention group will receive PEEP titrated using EIT with a stepwise decremental PEEP trial, while those in the control group will have PEEP set based on the FiO2-PEEP table. Other ventilator parameters will be managed according to the ARDSnet protocol.

The primary outcomes are blood oxygenation and pulmonary mechanics. Secondary outcomes include 28-day mortality, ventilator-free and shock-free days at 28 days, length of ICU and hospital stay, rate of successful weaning, the proportion requiring rescue therapies, complications, respiratory variables, and the Sequential Organ Failure Assessment (SOFA) score.

Before initiating recruitment maneuver, all patients were placed on mechanical ventilation set according to the ARDS network strategy for 10 minutes, ensuring SpO2 of 88-95%, PaO2 of 55-80 mmHg, and a mean arterial pressure (MAP) ≥ 65 mmHg.

* Patients received sedation and neuromuscular blockade to achieve full synchronization with the ventilator (RASS ≤ -3).
* The mode was set to Pressure-Controlled Ventilation (PCV): ΔP = 15 cmH2O, which was maintained constant during the recruitment maneuver, while FiO2, PEEP, and respiratory rate were kept as previously set.
* PEEP was incrementally increased by 5 cmH2O every minute: from 10 to 15, to 20, and finally to 25 cmH2O, with a maximum pressure limit of 40 cmH2O.
* Following the recruitment maneuver at the final PEEP level, the process of identifying the optimal PEEP was initiated.
* Then, PEEP will be set to 20 cmH2O and gradually decreased by 2 cmH2O every 30 seconds until it reached 6 cmH2O or SpO2 dropped to ≤ 80%.
* Selection of optimal PEEP: The optimal PEEP was defined as the intersection point between the alveolar overdistension and collapse curves as measured by the EIT system.

  * Termination Criteria: If persistent hypotension (mean arterial pressure decrease > 15 mmHg) or sustained hypoxemia (SpO2 < 85% for at least 1 minute) occurs during the recruitment maneuver maneuver, the procedure is terminated, and ventilator settings are returned to the parameters used prior to the recruitment maneuver.

Low FiO2 - PEEP table In the control group, patients set PEEP by low FiO2-PEEP table based on ARDSnet protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Intubated moderate and severe ARDS according to the New Global Definition (PaO2/FiO2 ≤200 mmHg).
* Used continuous sedation with or without paralysis.

Exclusion Criteria:

* Presence of pneumothorax that is either undrained or newly occurred.
* Unstable hemodynamics with a mean arterial pressure < 60 mmHg and unresponsive to resuscitation measures, and/or heart rate < 60 bpm.
* Contraindications for EIT (pacemakers, automatic external defibrillators, cases of chest trauma or recent chest surgery limiting EIT belt application).
* Pregnancy.
* Severe neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Oxygenation | at day 1, 2, 3, 4, 5, 6, 7
  PaO2/FiO2 will be evaluated via arterial blood gas analysis every day during the first week treatment.
Pulmonary Mechanic | at day 1, 2, 3, 4, 5, 6, 7
  Static Compliance

SECONDARY OUTCOMES:
Ventilator free days | up to 28 days
  Ventilator free days
Length of ICU stay | up to 28 days
  Days of ICU stay
Length of mechanical ventilated days | up to 28 days
  Days of received mechanical ventilation
Pneumothorax or barotrauma | up to 28 days
  new-onset of pneumothorax and barotrauma
Rescue therapies | up to 7 days
  Neuromuscular blocker, prone postition, ECMO
SOFA | at day 1, 3, 7
  Sequential Organ Failure Assessment
Mortality | up to 2 months
  the survival rate(survival/total) during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Center, Bach Mai Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Result] Jimenez JV, Weirauch AJ, Culter CA, Choi PJ, Hyzy RC. Electrical Impedance Tomography in Acute Respiratory Distress Syndrome Management. Crit Care Med. 2022 Aug 1;50(8):1210-1223. doi: 10.1097/CCM.0000000000005582. Epub 2022 May 23. PMID 35607967
- [Result] Matthay MA, Arabi Y, Arroliga AC, Bernard G, Bersten AD, Brochard LJ, Calfee CS, Combes A, Daniel BM, Ferguson ND, Gong MN, Gotts JE, Herridge MS, Laffey JG, Liu KD, Machado FR, Martin TR, McAuley DF, Mercat A, Moss M, Mularski RA, Pesenti A, Qiu H, Ramakrishnan N, Ranieri VM, Riviello ED, Rubin E, Slutsky AS, Thompson BT, Twagirumugabe T, Ware LB, Wick KD. A New Global Definition of Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2024 Jan 1;209(1):37-47. doi: 10.1164/rccm.202303-0558WS. PMID 37487152
- [Derived] Van Trung D, Giang BTH, Tuan DQ, Tan NC, Thach PT, Van Cuong B, Cuong NB, Anh TT, Anh NT, Van Huy N, Trieu HD, Van Trong N, Trang TT, Toan VX, Nam NH, Sam NT, Thanh TM, Dat NT, Hong NTP, Phuong PTH, Hien DD, Van Hoi D, Phong HT, Thu ND, Trang NT, Hieu NX, Dat HT, Phuong DX, Son DN. The impact of PEEP-guided electrical impedance tomography on oxygenation and respiratory mechanics in moderate-to-severe ARDS: a randomized controlled trial. Sci Rep. 2025 Nov 29;16(1):391. doi: 10.1038/s41598-025-29787-5. PMID 41318662